CLINICAL TRIAL: NCT01566006
Title: Mycophenolate Mofetil (MMF) ,Carnitine and Phosphodiesterase Type 5 Inhibitor, Three Potential Treatments for Resistant Proteinuria and for Slowing the Deterioration of Diabetic Nephropathy in Patients With Type II Diabetes Mellitus
Brief Title: Mycophenolate Mofetil, Carnitine and PDE5 Inhibitor, Three Potential Treatments for Resistant Proteinuria Slowing Diabetic Nephropathy Deterioration
Acronym: Myridian
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Nazareth Hospital, Israel (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, The Nazareth Hospital, Zaher armaly , M.D, Head of Nephrology Department, The Nazareth Hospital, Israel, The Nazareth Hospital, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nazh8827ctil
Record Dates: First submitted 2010-11-15; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Diabetic Nephropathy; Chronic Kidney Disease
Keywords: Mycophenolate mofetil (MMF); Diabetic Nephropathy; proteinuria; Diabetic Nephropathy in Chronic Kidney Disease patients stages 2-4
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Proteinuria | interventions — Mycophenolic Acid; Phosphodiesterase 5 Inhibitors; Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control group (No Intervention): group receiving the conventional treatment for DN
  Interventions: Drug: Mycophenolate Mofetil (MMF) ,phosphodiesterase 5 inhibitors , CARNITINE
- cellcept group (Experimental): additional to the conventional treatment patients will receive cellcept
  Interventions: Drug: Mycophenolate Mofetil (MMF) ,phosphodiesterase 5 inhibitors , CARNITINE
- carnitine group (Experimental): aside to the conventional treatment patients will receive carnitine
  Interventions: Drug: Mycophenolate Mofetil (MMF) ,phosphodiesterase 5 inhibitors , CARNITINE
- PDE5 group (Experimental): aside to the conventional treatment patients will receive PDE5 inhibitor
  Interventions: Drug: Mycophenolate Mofetil (MMF) ,phosphodiesterase 5 inhibitors , CARNITINE

INTERVENTIONS:
Drug: Mycophenolate Mofetil (MMF) ,phosphodiesterase 5 inhibitors , CARNITINE — effect of MMF on diabetic nephropathy patients by evaluating its effect on proteinuria and progression of kidney disease of diabetic origin

SUMMARY:
Diabetes mellitus (DM) is a growing disease and it is a public health concern, and projections of its future effect are alarming. About one third of those affected will develop diabetic nephropathy at 20 years after diagnosis. Of these patients, 20% will develop clinically end-stage renal disease ESRD, requiring renal replacement therapy (RRT). Patients with type 2 diabetes account for most patients with end stage renal disease (ESRD) and RRT.

To the best of the investigators knowledge, the effects of MMF on diabetic nephropathy in patients with DM type II were not studied so far. Therefore, the purpose of this pilot study is to evaluate the effects of Mofetil Mycophenolate (MMF) on proteinuria and progression of kidney disease of diabetic origin, in patients at high risk for progressive renal failure in whom other treatment modalities are insufficient or had failed.

DETAILED DESCRIPTION:
The pathophysiology of the diabetic nephropathy was initially considered to be merely secondary to a non-immune mechanism, specifically due to metabolic (hyperglycemia) and hemodynamic (glomerular capillary hypertension - mechanical stretching) factors. However, our understanding of the pathophysiological processes that lead to diabetic nephropathy and its progression is now clearer and involved not only a non immune mechanism, but also immune-mediated and inflammatory mechanism. Activation of the immune system, with the participation of a chronic inflammatory state, plays a central role in the pathogenesis of diabetic nephropathy. Evidence for the involvement of the immune system in the pathogenesis of diabetic nephropathy was derived from the elevated levels of proinflammatory cytokines such as IL-1, IL-6, IL-18, and TNF-α. These factors are important predictors of the development of diabetic nephropathy, and recently it was shown that these inflammatory cytokines play a determinant role in the development and progression of the microvascular diabetic nephropathy. The first published study that showed the implication of the inflammatory cytokines in the pathogenesis of the diabetic nephropathy was in 1991. Mycophenolate Mofetil (MMF) is an immunosuppressant drug, used to prevent rejection, especially acute rejection in various organ transplantations, mainly kidney transplantation since 1995. In the last decade there are increasing reports describing the beneficial use of MMF in immune- mediated and auto-immune disorders such as Systemic Lupus Erythematosus, IGA nephropathy and other glomerulopathies.

Unfortunately, the potentially beneficial effects of MMF on diabetic nephropathy were not examined in clinical DM and is limited to diabetic rats. In a recent study, Utimura et al. have demonstrated that MMF largely prevented the development of albuminuria and glomerular injury in experimental diabetic nephropathy. The beneficial effect of MMF was not related to its action on glomerular hemodynamic or improvement of metabolic control, but probably related directly to its immunosuppressive and anti-inflammatory properties.

ELIGIBILITY:
Inclusion Criteria:

1. T2 DM at age ≥18 y with at least 10 years duration of diabetes.
2. Proteinuria due to diabetic nephropathy of ≥ 2 gram/d treated with ACEi or ARBs at maximal tolerated dose or both of them.
3. CKD grade 1-3
4. Diabetic retinopathy (discuss with Zaid)

Exclusion Criteria:

1. Proteinuria of non diabetic origin
2. Overlap Proteinuria with diabetic nephropathy
3. Other intercurrent illness (fever due to infection ….) that can interfere with the urine protein secretion.
4. Acute Kidney Injury.
5. CKD stage 4-5.
6. New renoprotective treatment in the last 6 months before enrollment.
7. Changes in dosage of one of the renoprotective drugs in the last 6 months before enrollment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
proteinuria | before beginging of the treatment - baseline, after 1,2,3,4 weeks, after 1,2,3,4,5,6,7,8,9,10,11,12 months of the beginning of the treatment
  16 time points over 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Armaly, MD, Principal Investigator — Nazareth Hospital (E.M.M.S)
Locations (1):
- Nazareth hospital (EMMS), Nazareth, Israel